CLINICAL TRIAL: NCT04881318
Title: Compression Garments in the Community With POTS
Acronym: COM-COM-POTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: REB20-2224
Record Dates: First submitted 2021-04-29; First posted 2021-05-11 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Blood Pressure

STUDY DESIGN:
Intervention Model Description: This study will investigate the effects waist high compression garments and medications compared to waist-high compression garments and medications held. Participants will cross-over and complete both arms. If participants participate in the abdominal compression sub-study, the order of waist-high compression - abdominal compression will also be randomized.
Masking Description: It is not possible to mask participants to the compression garment intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Waist-High Compression Tights and Medications (Experimental): Participants will wear the waist-high compression garment while taking their regularly prescribed medications. This arm will evaluate the effects of waist-high compression garment treatment together with medications that modulate heart rate and blood pressure. This arm will also include control measurements before the garment is put on and after the garment is removed.
  Interventions: Other: Waist-High Compression Tights; Drug: Medications that modulate heart rate and blood pressure
- Waist-High Compression Tights and No Medications (Experimental): Participants will wear the waist-high compression garment while holding their regular medications that modulate heart rate and blood pressure (beta-blockers, midodrine, ivabradine, stimulants). This arm will look at the effectiveness of waist-high compression without medications. This arm will also include control measurements before the garment is put on and after the garment is removed.
  Interventions: Other: Waist-High Compression Tights
- Abdominal Compression Garments and Medications (Experimental): Participants will wear the abdominal compression garment while taking their regularly prescribed medications. This arm will evaluate the effects of abdominal compression garment treatment together with medications that modulate heart rate and blood pressure. This arm will also include control measurements before the garment is put on and after the garment is removed.
  Interventions: Other: Abdominal Compression Garments; Drug: Medications that modulate heart rate and blood pressure
- Abdominal Compression Garments and No Medications (Experimental): Participants will wear the abdominal compression garment while holding their regular medications that modulate heart rate and blood pressure (beta-blockers, midodrine, ivabradine, stimulants). This arm will look at the effectiveness of abdominal compression without medications. This arm will also include control measurements before the garment is put on and after the garment is removed.
  Interventions: Other: Abdominal Compression Garments

INTERVENTIONS:
Other: Waist-High Compression Tights — Waist-high compression tights providing 15-40 mmHg of pressure.
  Arms: Waist-High Compression Tights and Medications; Waist-High Compression Tights and No Medications
Other: Abdominal Compression Garments — Abdominal compression garment compressing the abdomen, buttocks, and upper thighs.
  Other Names: Abdominal shapewear, compression shorts
  Arms: Abdominal Compression Garments and Medications; Abdominal Compression Garments and No Medications
Drug: Medications that modulate heart rate and blood pressure — Medications that modulate heart rate and blood pressure that participants regularly take. These medications include beta-blockers, midodrine, ivabradine and stimulants.
  Arms: Abdominal Compression Garments and Medications; Waist-High Compression Tights and Medications

SUMMARY:
Compression Garments are a commonly prescribed treatment in Postural Orthostatic Tachycardia Syndrome (POTS). The effectiveness of a proof-of-concept compression garment has been demonstrated in an acute laboratory setting. It is not known if commercially available compression garments that participants wear in their every day lives are effective at improving heart rate and reducing symptoms in POTS. This trial will evaluate the use of commercially available waist-high and abdominal compression garments in adults diagnosed with POTS in a community setting.

DETAILED DESCRIPTION:
Current treatment of Postural Orthostatic Tachycardia Syndrome (POTS) involves pharmacological and non-pharmacological intervention including salt and fluid loading, exercise, physical countermanuevers, and compression garments. Lower extremity compression garments provide mechanical external pressure to the blood vessels in the legs, thighs and abdomen, shifting blood back to the central circulation to increase preload and stroke volume. With increased stroke volume, cardiac output is maintained without excessive tachycardia. Compression garments are commonly prescribed as a non-pharmacological treatment in POTS, but previously little evidence validated their use. A recent proof-of-concept compression garment study performed by our research lab demonstrated significant HR and symptom reductions with compression, with adult POTS patients in an acute laboratory setting. The effectiveness of commercially available compression garments in a community setting in POTS patients is not known.

In this study, the researchers will use commercially or medically (by prescription) available waist-high compression garments (WHC) that POTS patients use in their daily life, to evaluate compression as a viable long-term treatment option. Additionally, the researchers will perform an optional sub-study of abdominal compression garments (AC), evaluating their effectiveness. Results from this study will be used to inform the practicality and effectiveness of compression garments in the community setting. These findings could rapidly translate to the clinical setting and improve patient care.

Primary Hypothesis: Body compression with commercially available WHC will acutely reduce orthostatic tachycardia, when compared to no compression, in a community setting.

Sub-Study Hypothesis: Body compression with commercially available AC will acutely reduce orthostatic tachycardia, when compared to no compression, in a community setting.

The participant will complete the study in a community setting. The participant will be provided with the study supplies including a Holter monitor to wear during the study. The duration of the study will be up to 4 days in total. The "With Medications" phase is 2 days and the "Without Medications" phase is 2 days. The first randomization is whether to do the WHC studies first after medications have been held for at least 24h or without holding the medications. If the participant will be in the AC Sub-Studies, then they will do those studies during the same window of holding medications (or not) as the WHC study. The second randomization would determine the order of WHC-AC vs. AC-WHC during each window

For each study day, there will be a total of 4 standing tests. Participants will first put on the Holter monitor at the beginning of the study day. The first standing test (OVS #1) will be performed 30 minutes after the participant takes their medications but before putting on the compression garment. The participant will then put on the compression garment. The second (OVS #2) standing test will be performed 30 minutes after putting on the compression garment. The third (OVS #3) standing test will be performed a minimum of 3 hours after putting on the compression garment. After a minimum of 3hours, the participant will then remove the compression garment. The fourth standing test (OVS #4) will be performed 30 minutes after removing the garment. Participants will record their symptoms after each standing test, as well as medications taken each day in the provided study booklet.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of Postural Tachycardia Syndrome (POTS)
* Resident of Canada
* Owns waist-high compression garment: medical grade or commercially available tights with a pressure rating provided (e.g. 15-18 mmHg, 20-30 mmHg, 30-40 mmHg)
* Optional Sub-Study: owns an abdominal compression garment (e.g. abdominal shapewear, waist high shorts)
* Able to participate in a 4-day study (2x2 day segments with a 5-day washout period)

Exclusion Criteria:

* Overt cause for postural tachycardia (i.e., acute dehydration, thyroid disease) that precludes POTS diagnosis
* Not a resident of Canada
* Participants with somatization or severe anxiety symptoms will be excluded
* Pregnant (self-reported)
* Inability to tolerate compression garments for the duration of the study
* Does not own a waist-high compression garment
* Other factors which in the investigator's opinion would prevent the participant from completing the protocol, including poor compliance during previous studies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
WHC Heart Rate | 10 minutes
  The primary outcome is the delta HR (standing HR - supine HR) in orthostatic vital signs (OVS) #1 (prior to the WHC) and OVS #2 (30min after WHC is applied), in the "Without Medication" phase.
AC Heart Rate | 10 minutes
  The primary outcome is the delta HR (standing HR - supine HR) in orthostatic vital signs (OVS) #1 (prior to the AC) and OVS #2 (30min after AC is applied), in the "Without Medication" phase.

SECONDARY OUTCOMES:
Heart Rate - End of Study Day (WHC) | 10 minutes
  Delta HR measurement from OVS #3 (with WHC) compared to the delta HR from the OVS #4 (without WHC).
Heart Rate - WHC and Medication | 10 minutes
  The delta HR from OVS #1 - OVS #2 in the "With Medication" phase, compared to the delta HR from OVS #1 - OVS #2 in the "Without Medication" phase .
Heart Rate - WHC and AC | 10 minutes
  Delta HR from OVS #1 - OVS #2 on the WHC day, compared to OVS #1 - OVS #2 on the AC day, in the "With Medication" phase. This will provide an assessment of the differential efficacy of commercial WHC versus commercial AC in a home setting.
Heart Rate - End of Study Day (AC) | 10 minutes
  Delta HR measurement from OVS #3 (with AC) compared to the delta HR from the OVS #4 (without AC). This will provide an assessment of the efficacy of commercial AC with prolonged use during the day.
Heart Rate - AC and Medication | 10 minutes
  The delta HR from OVS #1 - OVS #2 in the "With Medication" phase, compared to the delta HR from OVS #1 - OVS #2 in the "Without Medication" phase. This will provide an assessment of the differential efficacy of commercial AC with and without POTS medications.

CONTACTS AND LOCATIONS:
Overall Officials: Satish M Raj, MD MSCI, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bourne KM, Karalasingham K, Siddiqui T, Mammarella B, Patel A, Exner DV, Sheldon RS, Raj SR. Abdominal-only Compression Garments Reduce Orthostatic Tachycardia and Improve Symptoms in Patients With Postural Orthostatic Tachycardia Syndrome. Can J Cardiol. 2025 Dec 1:S0828-282X(25)01481-3. doi: 10.1016/j.cjca.2025.11.038. Online ahead of print. PMID 41338488
- [Derived] Bourne KM, Karalasingham K, Siddiqui T, Patel A, Exner D, Sheldon R, Raj SR. A Community-Based Trial of Commercially Available Compression Tights in Patients With Postural Orthostatic Tachycardia Syndrome. JACC Clin Electrophysiol. 2025 Jan;11(1):179-190. doi: 10.1016/j.jacep.2024.09.033. Epub 2024 Nov 27. PMID 39614865